CLINICAL TRIAL: NCT01837849
Title: Comparative Effects of Recombinant Human Brain Natriuretic Peptide and Dobutamine on Acute Decompensated Heart Failure Patients With Different Blood BNP Levels
Brief Title: A Comparison of Recombinant Human Brain Natriuretic Peptide and Dobutamine
Status: Completed | Type: Observational
Sponsor: Nantong University (Other)
Responsible Party: Principal Investigator, Haiyan PAN, associate chief physician, Nantong University
Other Study IDs: AHNTU-2010-28
Record Dates: First submitted 2013-04-12; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Acute Decompensated Heart Failure
Keywords: heart failure; rhBNP; Dobutamine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To compare the therapeutic efficacy of recombinant human brain natriuretic peptide (rhBNP) with dobutamine on acute decompensated heart failure patients with different blood BNP levels

DETAILED DESCRIPTION:
Patients with acute decompensated heart failure (ADHF) whose left ventricular ejection fraction(LVEF) was <40%, were assigned to a high BNP group (BNP ≤ 3000 pg/mL) or an extra-high BNP group (BNP > 3000 pg/mL) , depending on their admission plasma BNP levels. Each group was then subdivided into rhBNP or dobutamine subgroups according to intravenous administration with either rhBNP or dobutamine for 24-72h. The effects of rhBNP and dobutamine on patients in the high and extra-high BNP groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* patients were classified as NYHA class III-IV
* ejection fraction <40%

Exclusion Criteria:

* intravenous administration with rhBNP or dobutamine in the 2 weeks before study entry
* acute myocardial infarction
* significant valvular stenosis
* serious ventricular arrhythmia (frequent ventricular premature beat of >5 bpm, nonsustained and sustained ventricular tachycardia)
* blood pressure <95/60 mmHg or >140/90 mmHg
* shock
* hypovolemia
* hepatic or renal impairment
* pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute decompensated heart failure who required hospitalization
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
left ventricular ejection fraction (LVEF) in the High and Extra-high BNP Groups | baseline and 5 days
Left ventricle end diastolic dimension (LVEDD)in the High and Extra-high BNP Groups | baseline and 5 days
Blood BNP in the High and Extra-high BNP Groups | baseline and 5 days

SECONDARY OUTCOMES:
Changes in New York Heart Association (NYHA) Class from Baseline to Day 5 after Treatment | baseline and 5 days
Blood Pressure (mmHg) | baseline and 5 days
Heart Rate | baseline and 5 days
Plasma Creatinine | baseline and 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Zhu, MD, Study Director — Affiliated Hospital of Nantong University

REFERENCES:
- [Derived] Pan HY, Zhu JH, Gu Y, Yu XH, Pan M, Niu HY. Comparative effects of recombinant human brain natriuretic peptide and dobutamine on acute decompensated heart failure patients with different blood BNP levels. BMC Cardiovasc Disord. 2014 Mar 4;14:31. doi: 10.1186/1471-2261-14-31. PMID 24593826